CLINICAL TRIAL: NCT07356479
Title: Enhancing Mental and Physical Health of Women Through Engagement and Retention (EMPOWER) 3.0 (QUE 25-015)
Brief Title: Enhancing Mental and Physical Health of Women Veterans 3.0
Acronym: EMPOWER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 26-001; 1I01RD000411-01A2 (Other Grant/Funding Number: VA Office of Research & Development)
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases; Overweight; Obesity; Hypertension; Cholesterol; Diabetes Mellitus; Prediabetic State; Menopause; Cognitive Behavioral Therapy; Primary Health Care; Stress Disorders, Post-Traumatic; Prevention; Implementation Science; Quality Improvement
Keywords: Cardiovascular diseases; Overweight; Obesity; Hypertension; Cholesterol; Diabetes Mellitus; Prediabetic State; Menopause; Cognitive Behavioral Therapy; Primary Health Care; Stress Disorders, Post-Traumatic; Prevention; Implementation science; Quality Improvement; Women; Veterans; Patient Participation; Patient Satisfaction; Patient Preference; Physicians, Primary Care; Physicians, Women; Health Behavior
MeSH Terms: conditions — Cardiovascular Diseases; Overweight; Obesity; Hypertension; Diabetes Mellitus; Prediabetic State; Stress Disorders, Post-Traumatic; Patient Participation; Patient Satisfaction; Patient Preference; Health Behavior

STUDY DESIGN:
Intervention Model Description: Cluster randomized type 3 hybrid implementation-effectiveness trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EBQI Booster (EBQI/B) (Active Comparator): A two-hour EBQI Booster delivered virtually to site-identified QI champions and local implementation teams for each EBP reviewing key EBQI components and providing examples grounded in the EBPs.
  Interventions: Behavioral: EBQI Booster (EBQI/B)
- EBQI Booster + External Facilitation (EBQI/B+EF) (Experimental): A two-hour EBQI Booster delivered virtually to site-identified QI champions and local implementation teams for each EBP reviewing key EBQI components and providing examples grounded in the EBPs, plus 12 months of external facilitation.
  Interventions: Behavioral: EBQI Booster + External Facilitation (EBQI/B+EF)

INTERVENTIONS:
Behavioral: EBQI Booster (EBQI/B) — EBQI is a systematic quality improvement method for engaging frontline practices in improvement that introduces "best science" and evidence in the service of operational goals. EBQI has been tested in several VA implementation trials and the VA Office of Women's Health (OWH) recently conducted a large-scale roll out of EBQI across VA women's health. Sites randomized to EBQI/B will receive a two-hour EBQI Booster delivered virtually to site-identified QI champions and local implementation teams for each EBP reviewing key EBQI components and providing examples grounded in the EBPs.
  Arms: EBQI Booster (EBQI/B)
Behavioral: EBQI Booster + External Facilitation (EBQI/B+EF) — EBQI is a systematic quality improvement method for engaging frontline practices in improvement that introduces "best science" and evidence in the service of operational goals. EBQI has been tested in several VA implementation trials and the VA Office of Women's Health (OWH) recently conducted a large-scale roll out of EBQI across VA women's health. External facilitation (EF) delivered by an expert facilitator from outside of the local implementation site, offers a supportive coaching process in which facilitators encourage interactive problem-solving in improvement efforts. EF is one of the most-studied implementation strategies. Sites randomized to EBQI/B+EF will receive a two-hour EBQI Booster delivered virtually to site-identified QI champions and local implementation teams for each EBP reviewing key EBQI components and providing examples grounded in the EBPs, plus 12 months of EF.
  Arms: EBQI Booster + External Facilitation (EBQI/B+EF)

SUMMARY:
Women Veterans are the fastest growing segment of VA users, with most users in midlife. This dramatic growth has created challenges for VA to ensure that appropriate services are available to meet women Veterans' needs, and that they will want and be able to use those services. Furthermore, few VA improvement efforts have focused on women Veterans' health and health care in midlife. The EMPOWER QUERI 3.0 Program is a cluster randomized type 3 hybrid implementation-effectiveness trial testing two strategies designed to support implementation and sustainment of evidence-based practices for women Veterans in at least 18 VA facilities from 4 regions.

DETAILED DESCRIPTION:
Women Veterans are the fastest growing group of Veterans Health Administration (VA) users. Of the 528,424 women Veterans who used VA care in FY19, nearly half were in midlife (aged 45-64). A growing number of studies identify gaps in health care for women Veterans in this life stage, during which menopause typically occurs, 49% of women Veterans meet criteria for obesity, and the risk of chronic disease increases dramatically. Furthermore, women Veterans have a high burden of trauma and physical and mental health comorbidities, which may exacerbate menopause symptoms and chronic disease risk as well as negatively impact healthcare engagement and trust. Notably, only 40% of women in VA care report "complete trust" in their VA provider. Lack of trust in VA can drive seeking community care, which is associated with lower quality of care, higher costs, and eventual attrition from VA. While VA has invested substantially in improving health care for women Veterans, continued improvement efforts are needed to ensure accessible, effective, trustworthy, and trauma-informed care for women Veterans, with concerted efforts for women in midlife.

The EMPOWER 3.0 Impact Goal is to optimize women Veterans' access to and quality and experience of care by offering trauma-informed, evidence-based interventions that meet high-priority health needs in midlife, and thereby, to increase women Veterans' trust, well-being, and engagement in VA care. This Impact Goal is guided by input from the investigators' longstanding VA operations partners: the Offices of Women's Health (OWH), Mental Health (OMH), Patient-Centered Care and Cultural Transformation (OPCC&CT), Rural Health (ORH), and the National Center for Health Promotion and Disease Prevention (NCP). To support sites with implementation, the investigators will leverage OWH's multi-year, multi-million dollar investment in rolling out Evidence-Based Quality Improvement (EBQI) across VA women's health. EBQI has demonstrated effectiveness in VA women's health, contributing to improved care services for women Veterans. In collaboration with OWH, the investigators' team now has a unique opportunity to assess the additional supports needed to successfully launch novel EBPs in women's health clinics across four partnering Veteran Integrated Service Networks (VISNs).

Specific Aims are to:

Aim 1. Support implementation and sustainment of three EBPs for women Veterans in midlife using an EBQI Booster (EBQI/B) strategy in 18 VA facilities that have completed the OWH EBQI initiative. Half of these sites (n=9) will be randomized to also receive 12 months of external facilitation (EF): EBQI/B+EF.

Aim 2. Conduct a multi-method implementation evaluation using a type 3 hybrid implementation-effectiveness cluster randomized trial design. The investigators will compare effectiveness of EBQI/B and EBQI/B+EF in terms of: (a) improved access to trauma-informed care for women Veterans; (b) implementation strategy fidelity, speed of implementation, and sustainment; (c) recipient perspectives on and experiences of EBP implementation; and (d) costs of implementation and business case analysis to support sustained EBP use.

Aim 3. Develop a translation-to-policy (T2P)-informed scale-up and evaluation plan to support sustainment, spread, and continuous improvement of trauma-informed EBPs in VA care.

The investigators will implement three EBPs: 1) Trauma-Informed Care (TIC), a VA-mandated set of activities and approaches that support trust and safety in primary care interactions, 2) Cognitive Behavioral Therapy for Symptoms of Menopause (CBT-SM), which provides group-based therapy, education, and personalized referrals for women across the menopausal transition; and 3) Women's MOVE!, which provides lifestyle and weight management support to enhance women Veterans' health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* This study is recruiting VA sites - not individual patients.
* Prior to randomization, the study team will work with sites to ensure they have met the preconditions necessary to enroll in the study, which includes VISN, regional and/or facility level leadership support for participation.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2030-09-30 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Engagement: TIC | 12 months
  # of women with shared decision-making treatment planning marker (1=WBS completed in EHR)
Engagement: CBT-SM | 12 months
  # women participating in CBT-SM (1=yes for one or more sessions)
Engagement: Women's MOVE! | 12 months
  # of women enrolled in Women's MOVE! (1=yes for one or more sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Alison B Hamilton, PhD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Melissa M Farmer Coste, PhD MS, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA; Bevanne A Bean-Mayberry, MD MHS, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Erin P Finley, PhD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Data sets underlying all publications resulting from the proposed research will not be shared outside VA, except as required under the Freedom of Information Act (FOIA), because VHA policy would prohibit re-disclosure.